CLINICAL TRIAL: NCT01685021
Title: A Phase IIa, Single-arm, Open-label Study of MOR00208, a Humanized Fc-Engineered Anti-CD19 Antibody, in Patients With Relapsed/Refractory B-cell Acute Lymphoblastic Leukemia (B-ALL)
Brief Title: Study of Fc-Optimized Anti-CD19 Antibody (MOR00208) to Treat B-cell Acute Lymphoblastic Leukemia(B-ALL)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: MorphoSys AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MOR208C202
Record Dates: First submitted 2012-09-03; First posted 2012-09-13 (Estimated); Results first posted 2018-02-22 (Actual); Last update posted 2018-02-22 (Actual); Status verified 2018-02

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: B-ALL; CD19; MOR208; MOR00208; Xmab5574; B-cell acute lymphoblastic leukemia; Fc-optimized Anti-CD19 Antibody
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma | interventions — tafasitamab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MOR00208 (formerly Xmab5574) (Experimental): intravenous Infusion of MOR00208, Fc-optimized Anti-CD19 Antibody
  Interventions: Drug: MOR00208 (formerly Xmab5574)

INTERVENTIONS:
Drug: MOR00208 (formerly Xmab5574)
  Other Names: MOR208

SUMMARY:
This is an open-label, multicentre study to characterize the safety and preliminary efficacy of the human anti CD19 antibody MOR00208 in adult subjects with relapsed/refractory B-cell acute lymphoblastic leukemia (B-ALL)

ELIGIBILITY:
Inclusion Criteria:

* Patients with previously treated Philadelphia-chromosome-negative B-ALL, with progression after at least one prior therapy. Patients with Philadelphia-chromosome-positive B-ALL can only be included if they are refractory or intolerant to at least one tyrosine-kinase-inhibitor.
* Male or female patients at least 16 years of age; if the patient is less than 18 years of age, the patient must have the ability to understand and give written assent in addition to the parent's/guardian's written informed consent.
* Patients with histologically confirmed diagnosis of B-ALL
* Mixed phenotype acute leukemia patients who have B cell immunophenotype.
* Patients with an Eastern Cooperative Oncology Group performance status of less than or equal to 2
* Patients with a total bilirubin of less than or equal to 2.0 mg/dL
* Patients with alanine aminotransferase or aspartate aminotransferase less than or equal to 2.5 times the upper limit of normal
* Patients with a creatinine level of less than or equal to 2.0 mg/dL
* If a female of childbearing potential, confirmation of a negative pregnancy test before enrollment and use of double-barrier contraception, confirmation of a negative pregnancy test before enrollment and use of oral contraceptive plus barrier contraceptive, or confirmation of having undergone clinically documented total hysterectomy, oophorectomy, or tubal ligation
* If a male, use of an effective barrier method of contraception during the study and for 3 months after the last dose if sexually active with a female of childbearing potential
* Patients with the ability to understand and give written informed consent and to comply with the study protocol

Exclusion Criteria:

* Patients who received previous treatment with an anti-CD19 antibody or fragments
* Receipt of anti-CD20 therapy no greater than 4 weeks before the first study dose
* Patients having undergone prior allogeneic stem cell transplantation within 3 months or having active graft versus host disease
* Patients with known hypersensitivity to any excipient contained in the drug formulation
* Patients with a New York Heart Association Class III or IV
* History of stroke or myocardial infarction within the last 6 months
* Patients with a history of positive human immunodeficiency virus test result (ELISA or western blot)
* Patients with positive hepatitis serology. Hepatitis B (HBV): Patients with positive serology for hepatitis B, defined as positive for hepatitis B surface antigen (HbsAg) or total anti-hepatitis B core antibody (anti-Hbc). Patients positive for anti- Hbc may be included if hepatitis B viral DNA is not detectable. Hepatitis C (HCV): Patients with positive hepatitis C serology (defined as positive for anti-hepatitis C virus antibody (anti-HCV) unless HCV-RNA is confirmed negative.
* Patients with active viral, bacterial, or systemic fungal infection requiring active parenteral treatment
* Patients who are receiving active treatment/chemotherapy for another primary malignancy or have received any treatment, including surgery, radiation, or chemotherapy, within the past 5 years (except ductal breast cancer in situ, for nonmelanoma skin cancer, prostate cancer not requiring treatment, and cervical carcinoma in situ)
* Patients who are pregnant or breastfeeding
* Patients with major surgery or radiation therapy within 4 weeks prior to first study dose

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2013-04; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elias Jabbour, MD, Principal Investigator — MDA; Rebecca Klisovic, MD, Principal Investigator — Ohio State University; Wing H. Leung, M.D., PhD, Principal Investigator — St. Jude Children's Research Hospital
Locations (3):
- United States (3):
  - Ohio State University Medical Center, Columbus, Ohio
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - University of Texas M.D. Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Derived] Klisovic RB, Leung WH, Brugger W, Dirnberger-Hertweck M, Winderlich M, Ambarkhane SV, Jabbour EJ. A phase 2a, single-arm, open-label study of tafasitamab, a humanized, Fc-modified, anti-CD19 antibody, in patients with relapsed/refractory B-precursor cell acute lymphoblastic leukemia. Cancer. 2021 Nov 15;127(22):4190-4197. doi: 10.1002/cncr.33796. Epub 2021 Aug 3. PMID 34343354

RESULTS

PARTICIPANT FLOW:
Groups:
- MOR00208 (Formerly Xmab5574): intravenous Infusion of MOR00208, Fc-optimized Anti-CD19 Antibody
  MOR00208 (formerly Xmab5574)
  Total Patients Screened: 30 Total patients Enrolled (at least one infusion with study treatment): 22
Period: Overall Study
Arm/Group | MOR00208 (Formerly Xmab5574)
Started | 22
Completed | 6 (Last patient last visit date. Study was Terminated prematurely.)
Not Completed | 16

BASELINE CHARACTERISTICS:
Groups:
- MOR00208 (Formerly Xmab5574): intravenous Infusion of MOR00208, Fc-optimized Anti-CD19 Antibody
  MOR00208 (formerly Xmab5574)
Arm/Group | MOR00208 (Formerly Xmab5574)
Number analyzed (Participants) | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.82 (17.098)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 12
Body Mass Index [Mean (Standard Deviation); unit: kg/m2] | 29 (8.496)

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: ORR= CR (Complete Remission) + PR (Partial Remission)
  Antitumor activity of MOR00208
Time Frame: Throughout during study until progression, after each treatment cycle
Measure: Number; unit: participants
Arm/Group | MOR00208 (Formerly Xmab5574)
Number analyzed (Participants) | 22
participants | 2

2. Secondary Outcome: Patients Response Duration Evaluation by Hematology, Bone Marrow Aspirates or Biopsy, CT
Description: Two patients had a response to treatment. For one of the two patients a progression was recorded, the other patient was censored due to an AE. Conse quently, the planned Kaplan-Meier analyses of response duration and time to hematological relapse could not be calculated.
Time Frame: Throughout during study until progression, after each treatment cycle
Measure: Number; unit: days
Arm/Group | MOR00208 (Formerly Xmab5574)
Number analyzed (Participants) | 22
days
  Responder 1 | 56
  Responder 2 | 28

3. Secondary Outcome: Safety Will be Evaluated by Assessing Adverse Events, Clinical Lab Data and Vital Signs, ECG, Physical Exam
Description: Number of patients with at least one treatment-emergent AE
Time Frame: weekly, up to 7 months
Measure: Number; unit: patients
Arm/Group | MOR00208 (Formerly Xmab5574)
Number analyzed (Participants) | 22
patients | 22

4. Secondary Outcome: Pharmacokinetics of MOR00208
Description: Steady State Trough Plasma Concentration (Cpre-dose) at 9th dose (infusion)
Time Frame: weekly, up to 16 weeks, based on samples taken Pre-dose (ie before infusion start)
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | MOR00208 (Formerly Xmab5574)
Number analyzed (Participants) | 22
mcg/mL | 198 (63.5)

5. Secondary Outcome: Number of Patients Who Develop Ant-MOR00208 Antibodies as a Measure of Immunogenicity
Time Frame: monthly, up to 7 months
Population: Anti-MOR208 antibodies were not observed in any patients treated during this study.
Measure: Number; unit: patients
Arm/Group | MOR00208 (Formerly Xmab5574)
Number analyzed (Participants) | 22
patients | 0

6. Secondary Outcome: Safety Will be Evaluated by Assessing Adverse Events, Clinical Lab Data and Vital Signs, ECG, Physical Exam
Description: Number of patients with treatment-emergent AEs
Time Frame: weekly, up to 7 months
Measure: Number; unit: number of patients with 1 or more AE
Arm/Group | MOR00208 (Formerly Xmab5574)
Number analyzed (Participants) | 22
number of patients with 1 or more AE | 22

ADVERSE EVENTS:
Time Frame: From signature of informed consent till up to 30 days after last study drug administration, or longer, as necessary.
Description: Treatment-related Adverse Events
Arm/Group | MOR00208 (Formerly Xmab5574)
All-Cause Mortality (participants affected / at risk) | 5/22
Serious Adverse Events (participants affected / at risk) | 17/22
Other Adverse Events (participants affected / at risk) | 22/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MOR00208 (Formerly Xmab5574) (N=22)
Disease Progression (General disorders) | 6 — SAEs occuring in more than 2 patients in the study
Pyrexia (General disorders) | 5 — SAEs occuring in more than 2 patients in the study
Febrile Neutropenia (Blood and lymphatic system disorders) | 4 — SAEs occuring in more than 2 patients in the study
Sepsis (Infections and infestations) | 3 — SAEs occuring in more than 2 patients in the study
Tumor lysis syndrome (General disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MOR00208 (Formerly Xmab5574) (N=22)
Infusion related reaction (General disorders) | 13
Fatigue (General disorders) | 9
Hypokalaemia (Metabolism and nutrition disorders) | 6
Constipation (Gastrointestinal disorders) | 6
Hyperglycaemia (Metabolism and nutrition disorders) | 6
Nausea (General disorders) | 6
Aspartate aminotransferase increased (Hepatobiliary disorders) | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5
Hyperkalaemia (Metabolism and nutrition disorders) | 5
Neutrophil count decreased (Blood and lymphatic system disorders) | 4
Abdominal pain (General disorders) | 4
Diarrhoea (Gastrointestinal disorders) | 4
Pyrexia (General disorders) | 4
Hypocalcaemia (Metabolism and nutrition disorders) | 4
Alanine aminotransferase increased (Hepatobiliary disorders) | 4
Anaemia (Blood and lymphatic system disorders) | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Platelet count decreased (Blood and lymphatic system disorders) | 4
Hypertension (Cardiac disorders) | 4
Gamma-glutamyltransferase increased (Hepatobiliary disorders) | 4
Hypomagnesaemia (Metabolism and nutrition disorders) | 4
Epistaxis (General disorders) | 3
Chills (General disorders) | 3
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3
Paraesthesia (Nervous system disorders) | 3
Oedema peripheral (General disorders) | 3
Headache (Nervous system disorders) | 3
Contusion (Injury, poisoning and procedural complications) | 3
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3
Confusional state (General disorders) | 3
Oedema (General disorders) | 3
White blood cell count decreased (Blood and lymphatic system disorders) | 2
Blood creatinine increased (Renal and urinary disorders) | 2
Pollakiuria (Renal and urinary disorders) | 2
Renal failure acute (Renal and urinary disorders) | 2
Hypotension (Vascular disorders) | 2
Vomiting (Gastrointestinal disorders) | 2
Agitation (General disorders) | 2
Dizziness (Nervous system disorders) | 2
Insomnia (Psychiatric disorders) | 2
Anxiety (Psychiatric disorders) | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 2
Presyncope (General disorders) | 2
Sinus tachycardia (Cardiac disorders) | 2
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2
Renal failure (Renal and urinary disorders) | 2
Mucosal inflammation (General disorders) | 2
Hyperuricaemia (Renal and urinary disorders) | 2
Ocular hyperaemia (Eye disorders) | 1
Blood albumin decreased (Investigations) | 1
Haematuria (Renal and urinary disorders) | 1
Blood amylase increased (Investigations) | 1
Blood glucose increased (Metabolism and nutrition disorders) | 1
Lymphopenia (Blood and lymphatic system disorders) | 1
Oral pain (General disorders) | 1
Chest discomfort (General disorders) | 1
Proctalgia (Gastrointestinal disorders) | 1
Decreased appetite (Gastrointestinal disorders) | 1
Cystitis (Renal and urinary disorders) | 1
Cytomegalovirus viraemia (Infections and infestations) | 1
Blood magnesium decreased (Metabolism and nutrition disorders) | 1
Graft versus host disease (Immune system disorders) | 1
Haemorrhoids (Gastrointestinal disorders) | 1
Hepatitis viral (Infections and infestations) | 1
Hepatorenal syndrome (Hepatobiliary disorders) | 1
International normalised ratio increased (Investigations) | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Lymphoedema (General disorders) | 1
Myalgia (General disorders) | 1
Sepsis (Infections and infestations) | 1
Tremor (General disorders) | 1
Urinary tract infection (Infections and infestations) | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1
Abdominal distension (General disorders) | 1
Dysgeusia (General disorders) | 1
Flushing (General disorders) | 1
Dysphonia (General disorders) | 1
Petechiae (Vascular disorders) | 1
Acidosis (Metabolism and nutrition disorders) | 1
Vision blurred (Eye disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Hyperhidrosis (General disorders) | 1
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1
Strabismus (Eye disorders) | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1
Device related infection (Infections and infestations) | 1
Weight increased (General disorders) | 1
Brachial plexopathy (Nervous system disorders) | 1
Malaise (General disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Syncope (Nervous system disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Migraine (General disorders) | 1
Lymph node pain (General disorders) | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1
Bradycardia (Cardiac disorders) | 1
Depression (Psychiatric disorders) | 1
Fall (Injury, poisoning and procedural complications) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Lung infection (Infections and infestations) | 1
Haemangioma of liver (Vascular disorders) | 1
Oropharyngeal pain (Gastrointestinal disorders) | 1
Tumour lysis syndrome (General disorders) | 1
Weight decreased (General disorders) | 1
Swelling face (General disorders) | 1
Gingival pain (Gastrointestinal disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Periodontal disease (Gastrointestinal disorders) | 1
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 1
Trigeminal nerve disorder (Nervous system disorders) | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Infection (Infections and infestations) | 1
Lethargy (General disorders) | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1
Pain in extremity (General disorders) | 1
Wound infection (Infections and infestations) | 1
Chest pain (Respiratory, thoracic and mediastinal disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Pharyngitis (Gastrointestinal disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Encephalopathy (Nervous system disorders) | 1
Dyskinesia (Nervous system disorders) | 1
Supraventricular tachycardia (Cardiac disorders) | 1
Blood alkaline phosphatase increased (Investigations) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 1
Asthenia (General disorders) | 1
Alpha haemolytic streptococcal infection (Infections and infestations) | 1
Corynebacterium infection (Infections and infestations) | 1
Lip disorder (Gastrointestinal disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Rash erythematous (Skin and subcutaneous tissue disorders) | 1
Hypoalbuminaemia (Investigations) | 1
Intracranial pressure increased (Nervous system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Allergic transfusion reaction (General disorders) | 1
Hyperphosphataemia (Metabolism and nutrition disorders) | 1
Leukaemic infiltration (General disorders) | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
As specified in the respective clinical trial agreements with the PI.